CLINICAL TRIAL: NCT03138681
Title: A Preliminary Clinical Study on the Rapid Antidepressant Effects of Adenosine Triphosphate (ATP) and Phosphocreatine Combinated With Fluoxetine
Brief Title: Rapid Antidepressant Effects of ATP and Phosphocreatine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-SJNK-001
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Adenosine Triphosphate; Phosphocreatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ATP (Experimental)
  Interventions: Drug: ATP
- phosphocreatine (Experimental)
  Interventions: Drug: Phosphocreatine

INTERVENTIONS:
Drug: Placebo — placebo is given intravenously twice a day for 14 days
  Arms: Placebo
Drug: ATP — ATP (100mg) is given intravenously twice a day for 14 days
  Arms: ATP
Drug: Phosphocreatine — Phosphocreatine (1g) is given intravenously twice a day for 14 days
  Arms: phosphocreatine

SUMMARY:
This is a preliminary, double-blind clinical trail aimed to investigate whether the combination of fluoxetine with ATP or phosphocreatine has a rapid antidepressant effect. 42 patients with major depressive disorder (Hamilton Depression Rating Scale (HAMD) score >= 20) will be recruited and divided into 3 groups randomly. This study involves two periods. In the first period, one group will be treated with fluoxetine and placebo, one with fluoxetine and ATP, and one with fluoxetine and phosphocreatine for 2 weeks. Placebo, ATP and phosphocreatine will be given intravenously, and fluoxetine orally. In the second period, each patient will be only given fluoxetine for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year-old male or female
* Major depressive disorder diagnosed by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Hamilton depression rating scale score >= 20 at screening
* Written informed consent

Exclusion Criteria:

* Participants of other clinical trials in recent 4 weeks
* Suicidal idea or action that requires hospitalization
* Post Traumatic Stress Syndrome in recent 6 months
* Secondary depression, or have a direct familial history of schizophrenia
* Diseases that prevent from appropriate expression of depressive emotion
* Psychiatric disorders including bipolar disorder and schizophrenia
* Severe heart, kidney, lung or liver diseases that require hospitalization
* Diabetes
* Neurologic disease (eg., epilepsy, infarct, multiple sclerosis, brain tumor)
* Inflammatory disease including autoimmune disease
* Taking anti-inflammatory medication
* Taking antiarrhythmic drugs, antidiabetic agents or tryptophan
* Substance abuse or dependence history in recent 6 months
* Pregnant or having plan to be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Hamilton depression rating scale during the first six weeks | baseline, 1st, 2nd, 4th, 6th week

SECONDARY OUTCOMES:
Changes in Patient Health Questionnaire (PHQ-9) during the first six weeks | baseline, 1st, 2nd, 4th, 6th week
Changes in Clinical global impression scale during the study | baseline, 2nd, 4th, 10th week
Side effects assessment during the first six weeks | 1st, 2nd, 4th, 6th week

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Cao X, Zang W, Tan S, Ou CQ, Shen X, Gao T, Zhao L. Intravenous administration of adenosine triphosphate and phosphocreatine combined with fluoxetine in major depressive disorder: protocol for a randomized, double-blind, placebo-controlled pilot study. Trials. 2019 Jan 9;20(1):34. doi: 10.1186/s13063-018-3115-4. PMID 30626424